CLINICAL TRIAL: NCT00112710
Title: A British Thoracic Oncology Group Phase III Trial of Gemcitabine Plus Cisplatin at 80mg/m Versus Gemcitabine Plus Carboplatin At 50 mg/m Versus Gemcitabine Plus Carboplatin AUC 6 in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine in Combination With Either Cisplatin or Carboplatin in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000429610; CRUK-BTOG2-LU3005; EU-20510
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether giving gemcitabine together with cisplatin is more effective than giving gemcitabine together with carboplatin in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying gemcitabine and cisplatin to see how well they work compared to gemcitabine and carboplatin in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of gemcitabine in combination with 2 different doses of cisplatin vs carboplatin, in terms of survival time, in patients with stage IIIB or IV non-small cell lung cancer.

Secondary

* Compare symptom control and quality of life of patients treated with these regimens.
* Compare response in patients treated with these regimens.
* Compare the dose intensity of these regimens in these patients.
* Compare the ratio of courses of treatment given as in-patient vs out-patient in these patients.
* Compare the intensity and number and duration of toxic episodes in patients treated with these regimens.
* Compare cost and cost-effectiveness of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to WHO performance status (0 vs 1 or 2), disease stage (IIIB vs IV), and participating center. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 1.
* Arm II: Patients receive gemcitabine as in arm I and cisplatin (at a lower dose than in arm I) IV over 1 hour on day 1.
* Arm III: Patients receive gemcitabine as in arm I and carboplatin IV over 1 hour on day 1.

In all arms, treatment repeats every 21 days for 2 courses. Patients are reassessed after 2 courses. Patients with responding disease or stable disease with symptom improvement receive 2 additional courses of therapy in the absence of disease progression or unacceptable toxicity. Patients with disease progression or stable disease without symptom improvement are removed from the study.

Quality of life is assessed at baseline, on day 1 of courses 2-4, at completion of study treatment, and then monthly for 6 months.

After completion of study treatment, patients are followed monthly for 6 months and then periodically thereafter for survival.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,350 patients (450 per treatment arm) will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following stage criteria:

  * Stage IIIB disease* that is not suitable for radical radiotherapy
  * Stage IV disease* NOTE: *Radiographically verified
* At least 1 measurable lesion by clinical examination or radiography
* No mixed histologies of small cell lung cancer and NSCLC
* No clinically apparent brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL

Hepatic

* AST < 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Alkaline phosphatase < 3 times ULN
* Bilirubin < 1.5 times ULN

Renal

* Creatinine clearance ≥ 60 mL/min (by Wright equation) OR ≥ 70 mL/min (by ^51Cr-EDTA clearance)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able and willing to participate in the quality of life assessment
* No pre-existing neuropathy > grade 2
* No other malignancy that would preclude study treatment or study comparisons
* No evidence of severe or uncontrolled systemic disease, significant clinical disorder, or laboratory finding that would preclude study participation
* No psychiatric disorder that would preclude study participation
* No other condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy, including neoadjuvant or adjuvant chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* No concurrent hormonal therapy except contraceptives or replacement steroids

Radiotherapy

* No prior radiotherapy

Surgery

* Recovered from prior surgery
* Prior surgical resection for NSCLC allowed

Other

* More than 12 weeks since prior investigational agents and recovered
* No other concurrent specific antitumor therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2005-03

PRIMARY OUTCOMES:
Length of survival

SECONDARY OUTCOMES:
Symptom control and quality of life as measured by the EORTC Quality of Life Questionnaire Core 30 Items and Lung Cancer supplement 13 together with EuroQol-5 domain questionnaire
Treatment response as measured by RECIST criteria
Dose intensity of chemotherapy
Ratio of treatment courses given as in-patient versus out-patient
Toxicity as measured by CTCAE v3.0
Treatment cost

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Jarrett, Study Chair — Institute of Clinical Research - Birmingham
Locations (2):
- United Kingdom (2):
  - Institute of Clinical Research - Birmingham, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England

REFERENCES:
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867
- [Derived] Ferry D, Billingham L, Jarrett H, Dunlop D, Woll PJ, Nicolson M, Shah R, Thompson J, Spicer J, Muthukumar D, Skailes G, Leonard P, Chetiyawardana AD, Wells P, Lewanski C, Crosse B, Hill M, Gaunt P, O'Byrne K. Carboplatin versus two doses of cisplatin in combination with gemcitabine in the treatment of advanced non-small-cell lung cancer: Results from a British Thoracic Oncology Group randomised phase III trial. Eur J Cancer. 2017 Sep;83:302-312. doi: 10.1016/j.ejca.2017.05.037. Epub 2017 Aug 4. PMID 28780466